CLINICAL TRIAL: NCT03784976
Title: Iyengar Yoga for Treatment of Endometriosis and Secondary Dysmenorrhea: A Randomized Controlled Clinical Trial
Brief Title: Iyengar Yoga Therapy for Dysmenorrhea and Endometriosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Kashif Ahmad, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18257
Record Dates: First submitted 2018-09-11; First posted 2018-12-24 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Secondary Dysmenorrhea; Dysmenorrhea; Dysmenorrhea Secondary; Polycystic Ovary Syndrome; Endometriosis; Fibroid; Menstrual Pain; Menstrual Disorder; Menstrual Discomfort
MeSH Terms: conditions — Dysmenorrhea; Polycystic Ovary Syndrome; Endometriosis; Leiomyoma; Menstruation Disturbances

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients in the intervention group will first undergo 3 months of regular care and then 3 months of biweekly yoga classes. Participants will complete surveys at baseline, 3 months (after of control care), 6 months (after 3 months of biweekly yoga classes), and 12 months (after 6 months of observation and optional yoga practice).
  Interventions: Other: Iyengar Yoga Therapy
- Control (No Intervention): The study lasts 12 months for the intervention and 9 months for the control group with an optional 3 month yoga therapy session offered at the end

INTERVENTIONS:
Other: Iyengar Yoga Therapy — 2 weekly yoga class (1.25 hours each)
  Other Names: Iyengar Yoga
  Arms: Intervention

SUMMARY:
The purpose of this clinical trial is to look at the effectiveness of prescribing yoga classes to patients with dysmenorrhea (irregular or painful periods), or other menstrual disorders on patients' self reported pain and quality of life.

Patients will be recruited from primary care clinics around Illinois, including Carle Hospital. This is a randomized trial in which patients will first be randomized into the control or intervention group. Patients in the control group will undergo usual care and be surveyed at baseline, 3 months, 6 months and 9 months. Patients in the control group will be offered the 3 months of yoga therapy complimentary after completing the 9 month control. Control patients who choose to participate in the yoga therapy will be asked to also complete the surveys at the end of the 3 month yoga intervention. Patients in the intervention group will first undergo 3 months of regular care and then 3 months of biweekly yoga classes. Participants will complete surveys at baseline, 3 months (after of control care), 6 months (after 3 months of biweekly yoga classes), 9 months, and 12 months (after 6 months of observation and optional yoga practice).

DETAILED DESCRIPTION:
Participants will contact the research team with the information on the flyer. Participants will be asked to come to the Iyengar Yoga Center (407 W Springfield Ave, Urbana, IL 61801) to receive more information. Participants will need to disclose their diagnosis to the research staff. If they are not aware of what their diagnosis is, they will need to contact their physician to get their official diagnosis. For example, a woman with dysmenorrhea may be diagnosed with poly cystic ovarian disease or endometriosis or idiopathic dysmenorrhea, or another reproductive disease; participants will need to know their specific diagnosis or find out their specific diagnosis and report it to the research staff. Participants can do this by calling their physicians. For participants that are unaware of their diagnosis, they may also request a copy of their medical records. These records may be shared with the research staff to help determine diagnosis. The research staff will not keep these medical records, but return them to the participants. Participants can then either consent on the first visit or choose to take time as much time as they need and return to the yoga center when they are ready to sign the consent form. Participants will complete the first round of surveys at the yoga center after they sign the consent form (20 minutes). Participants will receive an email or phone call from the study team to inform them of their randomization results.

A blind third party statistician will complete the randomization for all participants at the beginning of the study for all 90 participants and will email the study coordinator with the randomization results. Randomization will be done through a free online software called graphpad. (https://www.graphpad.com/quickcalcs/randomize1.cfm).

The study lasts 12 months for the intervention and 9 months for the control group with an optional 3 month yoga therapy session offered at the end: Once consented, participants will fill out baseline surveys, and then undergo 3 months of usual care (no intervention), the same baseline surveys will be filled out again, then participants will get biweekly free yoga therapy classes for 3 months, and surveys will again be completed at the end of the intervention. Patients will then have a 6 month follow up and will fill out the surveys one last time. Recruitment will occur on a rolling basis so patients may join the study at anytime and not have to wait for a batched group.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the proposed study is any menstruating female with dysmenorrhea, endometriosis, or any menstrual disorder. (Ages 12-65)

Exclusion Criteria:

* The exclusion criteria any one who has not reached menarche (age of menstruation) or who has reached menopause (no longer menstruates). This age range of exclusion is roughly defined as anyone younger than 12 and older than 65. Pregnant individuals are not eligible to participate in this study.

Ages: 12 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Must menstruate or be of menstruating age
Enrollment: 90 (Estimated)
Dates: Start 2018-07-03 (Actual); Primary Completion 2021-07-02 (Estimated); Study Completion 2021-07-02 (Estimated)

PRIMARY OUTCOMES:
NIH PROMIS Pain Interference Survey | baseline, 3 months, 6 months, 9 months, 12 months
  This survey is a 4 question short form. The PROMIS(r) Pain Interference instruments (adult and child) measure the self-reported consequences of pain on relevant aspects of a person's life and may include the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities.
NIH PROMIS Pain Intensity Survey | baseline, 3 months, 6 months, 9 months, 12 months
  This survey is a 3 question short form. The PROMIS Pain Intensity instrument assesses how much a person hurts.
NIH PROMIS Fatigue Survey | baseline, 3 months, 6 months, 9 months, 12 months
  This survey is a 4 question short form. The PROMIS Fatigue instruments evaluate a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles.
NIH PROMIS Physical Function Survey | baseline, 3 months, 6 months, 9 months, 12 months
  This survey is a 4 question short form. Physical Function measures self-reported capability rather than actual performance of physical activities. This includes the functioning of one's upper extremities (dexterity), lower extremities (walking or mobility), and central regions (neck, back), as well as instrumental activities of daily living, such as running errands.
NIH PROMIS Global Health Scale | baseline, 3 months, 6 months, 9 months, 12 months
  This survey is a 7 question short form. The PROMIS Global Health measures assess an individual's physical, mental, and social health.
Self-Reported Home Practice survey | baseline, 3 months, 6 months, 9 months, 12 months
  This survey is a 10 question survey about participants home yoga practice.
Menstrual Distress Questionnaire | baseline, 3 months, 6 months, 9 months, 12 months
  The Menstrual Distress Questionnaire (MDQ) is a standard method for measuring cyclical perimenstrual symptoms. It is used to help clinicians and researchers make systematic, empirical evaluations of a woman's symptoms, of treatments, and of etiological theories.
  The MDQ is a 46-item self-report inventory for use in the assessment and treatment of premenstrual and menstrual symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Iyengar Yoga Center, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF